CLINICAL TRIAL: NCT00935844
Title: An Open-Label, Dose Escalation, Phase I Study of TAK-901 in Adult Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Study of TAK-901 in Adults With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C19001
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: Advanced solid tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — TAK-901

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-901 Arm (Experimental)
  Interventions: Drug: TAK-901

INTERVENTIONS:
Drug: TAK-901 — This study consists of three sequential parts.
  Part 1: Escalating doses of TAK-901 will be administered via IV infusion over a 3-hour period on Days 1, 4, 8, 11, 15, and 18 of each 28-day cycle.
  Part 2: Escalating doses of TAK-901 (starting at one-third of the dose identified as the MTD in Part 1) will be administered as a 1-hour infusion on Days 1, 4, 8, 11, 15, and 18 of each 28-day cycle.
  Part 3: TAK-901 will be administered to approximately 20 patients using the dose identified as the MTD in the escalation phase. The infusion duration of TAK-901 will be determined after completion of Part 2.

SUMMARY:
This study is being conducted to evaluate the safety profile and the Maximum Tolerated Dose (MTD) of TAK-901 in adult patients with advanced solid tumors or lymphoma. This study will help to identify the recommended phase 2 dose and infusion duration, and describe the pharmacokinetics of TAK-901.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in the study:

* ECOG performance status of < or equal to 2.
* Diagnosis of solid tumor malignancy or lymphoma for which standard treatment is no longer effective.
* Have a radiographically or clinically evaluable tumor or lymphoma.
* Measurable disease as described in the protocol.
* Suitable venous access for the study-required blood sampling.
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse.
* Voluntary written consent.
* Weigh at least 45 kg.
* Recovered from the reversible effects of prior antineoplastic therapy.
* Meet clinical laboratory values during the screening period as specified in the protocol.
* Left ventricular ejection fraction (LVEF) > or equal to 50% by echocardiogram or multiple acquisition scan (MUGA).

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Diagnosis of primary CNS malignancy or carcinomatous meningitis.
* Patient has symptomatic brain metastasis.
* Prior bone allogeneic bone marrow or stem cell transplant.
* Prior radiotherapy involving > or equal to 30% of the hematopoietically active bone marrow, within 21 days before the start of the study drug.
* Systemic antineoplastic therapy within 28 days before the start of the study drug, except for luteinizing hormone-releasing-hormone (LHRH) agonist therapy.
* Exposure to nitrosureas or mitomycin C within 42 days before the start of the study drug.
* Treatment with monoclonal antibodies within 28 days before the start of the study drug.
* Known allergy or hypersensitivity to compounds of similar chemical composition to TAK-901 or its excipient, Captisol.
* Female patients who are lactating or who have a positive serum pregnancy test during the screening period or a positive serum pregnancy test during the screening period.
* Myocardial infarction within 6 months before enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Abnormalities on 12-lead electrocardiogram (ECG) as specified in the protocol.
* Infection requiring systemic anti-infective therapy within 14 days before the start of study drug.
* Known human immunodeficiency virus (HIV)positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Diagnosed or treated for another malignancy within 2 years before the start of study drug or previously diagnosed with another malignancy and have any evidence of residual disease.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment.
* Treatment with any investigational products within 28 days before the first dose of study drug.
* Systemic use of strong CYP3A inhibitors or inducers (as specified in the protocol) within 14 days before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To identify the MTD of TAK-901 administered as either a 3-hour or 1-hour infusion. | 12 months
To adaptively adjust the estimate of the MTD of TAK-901 from the escalation phase in an expansion cohort of subjects. | 12 months

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of TAK-901 and its primary metabolite (M-I). | 12 months
To evaluate disease response. | 12 months
To investigate the effect of TAK-901 on tumor proliferation. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - The University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Fox Chase Cancer Center, Rockledge, Pennsylvania